CLINICAL TRIAL: NCT05330962
Title: 10 Years Cardiovascular Risk Score Among Primary Health Care Centre Attendees, Assiut Governorate.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asma Ahmed Rafat Najeeb, registrar, Assiut University
Other Study IDs: Cardiovascular risk score
Record Dates: First submitted 2022-04-10; First posted 2022-04-15 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Cardiovascular Risk Score

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Framingham study cardiovascular disease 10-years risk assessment score — A personal interview questionnaire
  Other Names: ASCVD risk estimator

SUMMARY:
The study aim to assess cardiovascular risk score among patients of AlHadary primary health care centre in Waldeya, Assiut governorate. And to determine the awareness about cardiovascular risk among these patients as well.

DETAILED DESCRIPTION:
An analytical, cross-sectional study will be conducted in a primary health care center in Assiut governorate. Aiming to assess cardiovascular risk among attendees of the center and determine the awareness about cardiovascular risk among them.

ELIGIBILITY:
Inclusion Criteria:

* Male 30-65 years old, or female 40-70 years old.

Exclusion Criteria:

* History of ischemic heart disease, stroke, transitory ischemic attack (TIA) or peripheral artery disease (PAD) in electronic health record.
* History of diabetes

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Attendees of primary health care centre, Assiut governorate.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
The Framingham study cardiovascular disease 10 years risk assessment results | 1 year
  Participants will be categorized into four risk groups based on the 10 years ASCVD risk percentages.

SECONDARY OUTCOMES:
Total cardiovascular disease knowledge score results | 1 year
  will be calculated by summing the scores of respondents concerning cardiovascular disease types, heart attack symptoms, stroke symptoms and CVR factors. Total knowledge score will be 24. knowledge levels will be categorized as low knowledge, moderate knowledge and high knowledge.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yacoub M, Mayosi B, ElGuindy A, Carpentier A, Yusuf S. Eliminating acute rheumatic fever and rheumatic heart disease. Lancet. 2017 Jul 15;390(10091):212-213. doi: 10.1016/S0140-6736(17)31608-2. No abstract available. PMID 28721865
- See also: Importance of Lifestyle Modification on Cardiovascular Risk Reduction COUNSELING STRATEGIES TO MAXIMIZE PATIENT OUTCOMES — https://journals.lww.com/jcrjournal/Fulltext/2020/05000/Importance_of_Lifestyle_Modification_on.2.aspx?context=LatestArticles
- See also: Cardiovascular Risk Awareness and Calculated 10-Year Risk Among Female Employees at Taibah University 2019 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8520983/